CLINICAL TRIAL: NCT05431257
Title: Phase II Study of Azacitidine in Combination With Low Dose Intensity Venetoclax in Patients With Acute Myeloid Leukemia With Integration of Explorative Multi-omics and ex Vivo Drug Screening Data
Brief Title: Azacitidine in Combination With Low Dose Intensity Venetoclax in Patients With AML Incl. Explorative AML Profiling
Acronym: LD-VenEx
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Helse Stavanger HF (Other Government); University Hospital of North Norway (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other); Vestre Viken Hospital Trust (Other); Helse Møre og Romsdal HF (Other Government); Karolinska University Hospital (Other); Skane University Hospital (Other); Uppsala University Hospital (Other); Helsinki University Central Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Kim Theilgaard-Mönch, MD, DMSc, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21030117
Record Dates: First submitted 2022-06-01; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elderly/unfit AML patients or sec. and R/R AML patients (Experimental)
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Standard azacytidine treatment (AZA; D1-D7, 75mg/m2 qd) in combination with a short duration of "low-dose" venetoclax treatment (LD-VEN; D1-D14 before CR and D1-D7 after CR, 400mg qd) per 28 days cycle for elderly/unfit (arm 1) and relapsed/refractory (arm 2) patients with acute myeloid leukemia.

SUMMARY:
Multi-center phase II study of standard azacytidine treatment (AZA; D1-D7, 75mg/m2 qd) in combination with a short duration of "low-dose" venetoclax treatment (LD-VEN; D1-D14 before CR and D1-D7 after CR, 400mg qd) per 28 days cycle for elderly/unfit (arm 1) and relapsed/refractory (arm 2) patients with acute myeloid leukemia.

AZA and LD-VEN treatment is combined with exploratory AML profiling using established platforms for OMICs analyses and ex vivo drug sensitivity and resistance testing. This will validate the feasibility of AML profiling in a clinical setting to predict responders and non-responders to AZA/LD-VEN therapy. The exploratory AML profiling program will also identify biomarkers as well as novel drugs and drug combinations applicable for treatment of AML patients in future clinical trial initiatives.

DETAILED DESCRIPTION:
Multi-center phase II study of standard azacytidine treatment (AZA; D1-D7, 75mg/m2 qd) in combination with a short duration of "low-dose" venetoclax treatment (LD-VEN; D1-D14 before CR and D1-D7 after CR, 400mg qd) per 28 days cycle for elderly/unfit (arm 1) and relapsed/refractory (arm 2) patients with acute myeloid leukemia.

AML patients will be subjected to conventional diagnostic workup to assess if they fulfil eligibility criteria. As part of the exploratory trial program, bone marrow (BM) and peripheral blood (PB) samples will be subjected to functional AML profiling including OMICs analyses and immediate ex vivo drug sensitivity and resistance testing (DSRT). The treatment period with AZA/LD-VEN begins after completion of the diagnostic workup period, and includes drug treatment, clinical assessment, QoL assessment, and analysis of relevant follow-up BM and PB samples according to a detailed study event schedule. Patients will receive repeated cycles of treatment with AZA (D1-D7, 75mg/m2 qd) in combination with LD-VEN (D1-D14 before CR and D1-D7 after CR, 400mg qd) every 4 weeks. Patients exhibiting clinical response will continue treatment with AZA/LD-VEN for a maximum of two years or until withdrawal of consent, disease progression, unacceptable toxicity, intolerance, lack of compliance, unresponsiveness after three cycles of study treatment, or if they obtain CR and proceed to allogeneic stem cell transplantation. Clinical response (CR/CRi/MLFS=morphologic leukemia-free state/PR=partial remission), survival information (OS/DOR=duration of response/EFS=event-free survival), and QoL data will be collected for all patients independently on their response to AZA/LD-VEN treatment. Survival information and post-treatment follow-up (i.e. all post-treatment AML therapies including dates of initiation and completion, the date and cause of death) will be collected every three months for the first two years and thereafter annually for the following three years after End-Of-Treatment or withdrawal from study treatment, or until death of the patient.

The exploratory program will validate the feasibility of comprehensive OMICs profiling and ex vivo drug sensitivity and resistance testing in a clinical setting to predict responders and non-responders to AZA/LD-VEN therapy. The exploratory AML profiling program is expected to identify biomarkers as well as novel drugs and drug combinations applicable for treatment of AML patients that are refractory or suffer from relapse after AZA/LD-VEN treatment in future clinical trial initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients who present with one of the following (except acute promyelocytic leukemia).

  1. De novo or secondary AML unfit for standard induction therapy
  2. Relapsed/refractory AML after at least 1 line of prior therapies
* Written informed consent to participate in an exploratory research protocol including bio-banking, comprehensive AML profiling (genomics, transcriptomics, proteomics, etc.) and ex vivo drug sensitivity testing to assess venetoclax and other drug sensitivities.

  a) All patients are treated with azacitidine+venetoclax irrespective of the ex vivo screening results.
* ECOG Performance status ≤ 2 for patients ≥ 75 years of age OR ≤ 3 for patients ≥ 18 to 74 years of age.
* Leukocyte count < 25 x10E9/l. Hydroxyurea use is permitted to meet this criterion
* Adequate renal function as demonstrated by a calculated creatinine clearance ≥ 30 mL/min; determined by the Cockcroft Gault formula.
* Adequate liver function as demonstrated by

  1. alanine aminotransferase (ALT) ≤ 4.0 × ULN.
  2. bilirubin ≤ 1.5 × ULN.
* Specific inclusion criteria for elderly/unfit AML patients:

  1. ≥ 70 years of age OR
  2. ≥ 18 to 69 years of age and ineligible for intensive chemotherapy meeting at least one of the following criteria:

     * Clinically significant comorbidities, as reflected by at least 1 of the following criteria:

       * Left ventricular ejection fraction (LVEF) < 50%.
       * Lung diffusion capacity for carbon monoxide (DLCO) ≤ 65% of expected.
       * Forced expiratory volume in 1 second (FEV1) ≤ 65% of expected.
       * Chronic stable angina or congestive heart failure controlled with medication.
       * Alanine aminotransferase (ALT) 3.0-4.0 × ULN.
     * Other contraindication(s) to anthracycline therapy (must be documented).
     * Adverse risk genetics (ELN criteria) associated with poor outcome with standard chemotherapy.
     * Patient declines intensive chemotherapy.
     * Secondary AML after previous disease modifying treatment (i.e. HMA/induction chemotherapy and/or allogeneic stem cell transplantation) of clonal myeloid diseases such as MDS, MDS/MPN, or MPN.
* Specific inclusion criteria for relapsed AML patients:

  1. ≥ 55 years of age with non-CBF AML relapse OR
  2. ≥ 18 of age and meeting at least one of the following criteria:

     * Not candidate for intensive chemotherapy (see criterion 8).
     * Relapse after chemotherapy, or monotherapy with HMA, or allogeneic stem cell transplantation. (note: patients with 4th or higher relapse are excluded).
     * Patient declines intensive chemotherapy.
* Specific inclusion criteria for refractory AML patients:

Patients who fail to achieve a complete or partial remission after previous monotherapy with HMA or induction chemotherapy (at least 1 cycle of chemotherapy containing cytarabine or clofarabine, in combination with a topoisomerase II inhibitor (e.g. anthracycline or mitoxantrone).

Exclusion Criteria:

* Acute promyelocytic leukemia (APL).
* Patients with 4th or higher AML relapse.
* Leukemic cell content (blast percentage) in bone marrow/peripheral blood < 10 %.
* ECOG >3.
* Prior venetoclax treatment for myeloid malignancy.
* AML patients with CNS involvement (note: cerebrospinal fluid or radiological investigations are not required without clinical suspicion).
* HIV infection or active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection that is not controlled with antiviral medication with the definition hereof at the discretion of the investigator.
* Cardiovascular disability status of New York Heart Association Class ≥ 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in palpitations, fatigue, dyspnea, or anginal pain.
* Evidence of clinically significant condition(s), which at the investigator's discretion would adversely affect the patient's participation in this study (including but not limited to):

  1. Chronic respiratory disease that requires continuous oxygen use.
  2. Systemic uncontrolled infection requiring therapy (viral, bacterial or fungal).
  3. Malabsorption syndrome or other condition that precludes enteral route of administration.
  4. Uncontrolled GVHD.
* Previous malignancies with the exception of previous malignancy treated successfully with curative intent and indolent/smoldering malignancies (defined at the investigator's discretion).
* Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment).
* Fertile men or women of childbearing potential unless:

  1. Surgically sterile or ≥ 2 years after the onset of menopause.
  2. Willing to use two methods of reliable contraception including one highly effective contraceptive method (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 3 months after the end of study treatment.
* Known hypersensitivity to venetoclax or azacitidine or excipients of any of the drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1-1,5 year
  ORR(%) = CR rate(%)+CRi rate(%)+MLFS(%)
Composite complete remission rate | 1-1,5 year
  Composite CR rate (%) = CR rate (%) + CRh rate (%)
Partial remission rate | 1-1,5 year
  PR rate (%)

SECONDARY OUTCOMES:
Overall survival | 3,5-5 years
  Overall survival (OS) (months)
Duration of response | 3,5-5 years
  Duration of response (DOR) (months)
Event free survival | 3,5-5 years
  Event free survival (EFS) (months)
Frequency and severity of adverse events | 3-3,5 years
  Frequency and severity of adverse events (hematologic toxicities-AE grade 3+4, febrile neutropenia, days until neutrophil recovery ≥ 0.5 x 10E9/l and platelet recovery ≥ 50 x 10E9/l, severe AE grade 3+4).
The correlation of ex vivo drug sensitivity with specific clinical responses | 1,5-2 years
  The correlation of ex vivo drug sensitivity with specific clinical responses (OS, DOR, EFS, MRD status).
The correlation of venetoclax blood concentrations with specific responses | 1,5-2 years
  The correlation of venetoclax blood concentrations with specific responses (OS, DOR, EFS, MRD status).
Quality-of-Life | 3-3,5 years
  Quality-of-Life (QoL) as assessed by European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire - C30 (EORTC-QLQ-C30), including domains and scale 1-4 - (1) Not at all, (2) a little, (3) quite a bit, (4) very much.
Quality-of-Life | 3-3,5 years
  Quality-of-Life (QoL) as assessed by European Quality-of-Life - 5 Dimensions - 5 Level (EQ-5D-5L) questionnaire, including EQ-5D domains and visual analogue scale (VAS score 0-100).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No